CLINICAL TRIAL: NCT03897257
Title: A Multicenter, Randomized, Double-Blinded, Parallel Group Comparison Study of the Safety and Efficacy of UHE-103 in Subjects With Moccasin-Type Tinea Pedis
Brief Title: A Comparison Study of UHE-103 Cream in Subjects With Moccasin Type Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 146-9252-201
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Intervention Model Description: Five Arms:
  * 3 Arms of Monotherapy : UHE-103A1 cream (Drug A low dose concentration) or UHE-103A2 cream (Drug A high concentration) or UHE-103B cream (Drug B comparator)
  * 2 Arms of combination therapy: UHE-103A1B cream (Drug A low dose + Drug B), or UHE-103A2B cream (Drug A high dose + Drug B)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- UHE-103A1 cream (Experimental): Topical cream applied twice daily for 2 weeks.
  Interventions: Drug: UHE-103A1 cream
- UHE-103A2 cream (Experimental): Topical cream applied twice daily for 2 weeks.
  Interventions: Drug: UHE-103A2 cream
- UHE-103B cream (Experimental): Topical cream applied twice daily for 2 weeks.
  Interventions: Drug: UHE-103B cream
- UHE-103A1B cream (Experimental): Topical cream applied twice daily for 2 weeks.
  Interventions: Drug: UHE-103A1B cream
- UHE-103A2B cream (Experimental): Topical cream applied twice daily for 2 weeks.
  Interventions: Drug: UHE-103A2B cream

INTERVENTIONS:
Drug: UHE-103A1 cream — Investigational mono-therapy cream (containing drug A [low dose]). Drug A is an antifungal agent.
  Arms: UHE-103A1 cream
Drug: UHE-103A2 cream — Investigational mono-therapy cream (containing drug A [low dose]). Drug A is an antifungal agent.
  Arms: UHE-103A2 cream
Drug: UHE-103B cream — Comparator mono-therapy cream (containing drug B). Drug B is a keratolytic agent.
  Arms: UHE-103B cream
Drug: UHE-103A1B cream — Investigational combination-therapy cream (containing drug A [low dose antifungal] + drug B [keratolytic]).
  Arms: UHE-103A1B cream
Drug: UHE-103A2B cream — Investigational combination-therapy cream (containing drug A [high dose antifungal] + drug B [keratolytic]).
  Arms: UHE-103A2B cream

SUMMARY:
The study is being done to determine and compare the safety and effectiveness of an investigational combination therapy (low and high concentrations) versus mono-therapy (low and high concentrations) or mono-therapy (fixed concentration) in subjects with moccasin type tinea pedis.

DETAILED DESCRIPTION:
UHE-103 cream is an investigational combination drug to treat moccasin type tinea pedis, a fungal infection that affects the feet and toes. Eligible subjects will be assigned to one of the 5 possible treatment groups and participate for a total of 6 weeks. Subjects will apply their assigned test drug twice daily for 2 weeks. Each subject will then be assessed for safety and efficacy at week 4 and week 6. There will be a total of 5 clinic visits: 1 screening/baseline visit (Day 1), 2 treatment visits (Days 8 and 15), and 2 follow-up visits (Days 29 and 43).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female, 16 years of age or older.
* Clinical diagnosis of moccasin type tinea pedis
* Microscopic evidence (positive KOH) of the presence of fungi
* Provided written informed consent/assent
* In general good health

Exclusion Criteria:

* Pregnant or lactating or planning to get pregnant while on the study
* Has concurrent tinea infection (e.g., tinea versicolor, tinea cruris)
* Other skin disease which might interfere with the evaluation of tinea pedis
* History of diabetes mellitus or is immunocompromised
* Currently enrolled in an investigational drug or device study
* Used an investigational drug or investigational device treatment within 30 days prior to Visit 1 (Study Day 1)/Baseline

Other protocol defined inclusion or exclusion criteria assessed by the study staff may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Complete Cure at End of Study | Day 43
  Proportion of subjects with Complete Cure (negative fungal test & no clinical disease-induced signs and symptoms) at end of study (EOS).

SECONDARY OUTCOMES:
Effective treatment | Day 43
  Proportion of subjects with Effective Treatment (negative fungal test & no to mild clinical disease-induced signs and symptoms) at EOS.
Mycological Cure | Day 43
  Proportion of subjects with Mycological Cure (negative fungal test) at EOS.

CONTACTS AND LOCATIONS:
Overall Officials: Marietta Radona, MD, Principal Investigator — Therapeutics, Inc.
Locations (12):
- United States (11):
  - Site 03, San Diego, California
  - Site 12, Melbourne, Florida
  - Site 06, Miami, Florida
  - Site 09, North Miami Beach, Florida
  - Site 07, Rolling Meadows, Illinois
  - Site 11, Fridley, Minnesota
  - Site 04, Rochester, New York
  - Site 01, Austin, Texas
  - Site 02, Houston, Texas
  - Site 10, San Antonio, Texas
  - Site 05, Norfolk, Virginia
- Site 08, Cidra, Puerto Rico

IPD SHARING:
Plan to Share IPD: No